CLINICAL TRIAL: NCT07181070
Title: The Use of Indocyanine Green Fluorescence (ICG) During Laparoscopic Heller- Dor: a Prospective Study
Brief Title: The Use of Indocyanine Green Fluorescence (ICG) During Laparoscopic Heller- Dor
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe Palomba, Principal Investigator, Federico II University
Other Study IDs: 09082022
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Achalasia, Esophageal; Achalasia; Indocyanine Green (ICG); Indocyanine Green
Keywords: achalasia; Laparoscopic Heller-Dor; Indocyanine Green Fluorescence
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard group: IGC group

SUMMARY:
The aim this prospective observational study is to evaluate the role of Indocyanine Green Fluorescence (ICG) in patients with achalasia underwent to Heller-Dor laparoscopic. The main gol are:

* If with use of ICG iatrogenic mucosal leaks can be identified and, if necessary, improve the myotomy.
* Assess the need for postoperative radiographic control using esophagogastric radiography with gastrografin.
* Compare clinical characteristics, perioperative outcomes, and 12-month postoperative follow-up between the two populations.

DETAILED DESCRIPTION:
Achalasia is a rare disease of motility characterized by dysfunction of low esophageal sphincter (LES). This disease is divided according to Chicago classification. Laparoscopic Heller - Dor is gold standard of types I and II Achalasia. The use of intraoperative indocyanine green (ICG) fluorescence in recent years is becoming an interesting and innovative tool for surgical procedures. Its use is widely described in surgery The aim of our study is to value the role of ICG for this surgery. The investigators prospectively enrolled achalasic patients undergoing laparoscopic Heller -Dor .

ELIGIBILITY:
Inclusion Criteria:

* patients with achalasia of type I and II
* patients undergoing laparoscopic Heller-Dor
* patients older than 18 years

Exclusion Criteria:

* Patients <18 years of age;
* Uncooperative patients and/or patients unable to provide informed consent
* ASA ≥4
* BMI ≥30
* Patients previously treated with other endoscopic/surgical procedures (botulinum toxin injections, dilation, POEM, myotomy)
* Patients with achalasia type III
* Patients with megaesophagus
* Allergy to dyes or contrast agents included in the protocol (e.g., indocyanine green, barium, gastrografin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient has type I or type II esophageal achalasia and was treated with the Heller-Dor laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
mucosal leak | Intraoperative
  Directly visualize intraoperatively the presence or absence of an esophageal mucosal lesion through the color change due to indocyanine green fluorescence.
Completeness of myotomy | intraoperative
  Intraoperatively visualize the presence or absence of residual muscle fibers after myotomy through the use of indocyanine green fluorescence.

SECONDARY OUTCOMES:
Length of stay | From the first to the fourth post-operative day
  days of hospitalization from first postoperative day to discarge
Perioperative complications | Perioperative/Periprocedural
  Based on Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Aprea, Prof., Study Director — Federico II University
Locations (1):
- Università degli Studi di Napoli, Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Romanzi A, D'Alba L, Campagna P, Mancini R, Pernazza G. Robotic Heller-Dor procedure for oesophageal achalasia: Fluorescence-guided intraoperative assessment of myotomy. A retrospective single-centre experience. Int J Med Robot. 2022 Aug;18(4):e2411. doi: 10.1002/rcs.2411. Epub 2022 May 4. PMID 35472736
- [Background] Patel J, Kalikar V, Patankar R, Supe A. Is Indocyanine Green the New Gold Standard for Checking Completion of Laparoscopic Heller's Cardiomyotomy? Cureus. 2024 Dec 8;16(12):e75344. doi: 10.7759/cureus.75344. eCollection 2024 Dec. PMID 39781145
- [Background] Palomba G, Basile R, Capuano M, Pesce M, Rurgo S, Sarnelli G, De Palma GD, Aprea G. Nasogastric tube after laparoscopic Heller-Dor surgery: Do you really need it? Curr Probl Surg. 2024 Apr;61(4):101457. doi: 10.1016/j.cpsurg.2024.101457. Epub 2024 Feb 15. No abstract available. PMID 38548426